CLINICAL TRIAL: NCT03980028
Title: Role of Surgery in Advanced Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Institut Bergonié (Other); Institut Paoli-Calmettes (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Hospital Universitario La Paz (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: 18 HLGENF 01
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Cancer
Keywords: surgery; cancer; ovarian; advanced
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To demonstrate that ultra-radical surgery with multiple visceral resections and high tumor burden prior to surgery independently reduces the survival of patients with advanced ovarian cancer treated with complete cytoreductive surgery.

DETAILED DESCRIPTION:
Primary objective :

To demonstrate that ultra-radical surgery with multiple visceral resections and high tumor burden prior to surgery independently reduces the survival of patients with advanced ovarian cancer treated with complete cytoreductive surgery.

Secondary objectives:

1. Demonstrate that, in patients with advanced ovarian cancer (FIGO stage IIIC-IVB) treated by complete cytoreduction surgery, the high tumor load before surgery decreases survival. / Evaluate whether there is a sub-group of patients at risk for whom the high tumor burden prior to surgery reduces survival.
2. Demonstrate that, in patients with advanced ovarian cancer (FIGO stage IIIC-IVB) treated by complete cytoreduction surgery, the extension of carcinomatosis to the upper abdomen reduces the chances of survival. / Assess whether there is a subgroup of patients at risk for whom the extension of carcinomatosis to the upper abdomen reduces survival.
3. Demonstrate that, in patients with advanced ovarian cancer (FIGO Stage IIIC-IVB) treated by complete cytoreduction surgery, invasion of the celiac lymph nodes reduces survival rates. / Assess whether there is a subset of patients at risk where the invasion of the celiac lymph nodes reduces survival.
4. Demonstrate that, in patients with advanced ovarian cancer (FIGO stage IIIC-IVB) treated with complete cytoreduction surgery, combination with surgical procedures reduces survival. / Evaluate whether there is a sub-group of at-risk patients for whom the combination of surgical procedures with ultra-radical surgery reduces survival.

ELIGIBILITY:
Inclusion Criteria:

* confirmed histological diagnosis of ovarian epithelial cancer
* complete cytoreduction surgery

Exclusion Criteria:

* women under 18 years or presence of residual tumor >2.5mm after surgery or lack of data on performed surgical procedures or surgery performed before 2008, January or after 2015, Decembrer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ovarian cancer
Study Population: patients diagnosed with advanced epithelial ovarian cancer (IIIC-IVB of FIGO 2014) treated with cytoreduction surgery between 2008, January and 2015, December
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Patient survival | 4 years
  patient survival after surgery (patient record)
Evaluation of the tumor burden | 1 day
  Measurement of tumor size before surgery (patient record)

SECONDARY OUTCOMES:
Evaluation of the extension of carcinomatosis | 1 day
  Number of tumor nodules before surgery (patient record)
Evaluation of the invasion of celiac lymph nodes | 1 day
  Number of celiac lymph nodes before surgery (patient record)
Combination of surgical procedures | 1 day
  Number and type of combination of surgical procedures (patient record)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius Regaud - IUCT-Oncopole, Toulouse, Occitanie, France

REFERENCES:
- [Result] Bristow RE, Chi DS. Platinum-based neoadjuvant chemotherapy and interval surgical cytoreduction for advanced ovarian cancer: a meta-analysis. Gynecol Oncol. 2006 Dec;103(3):1070-6. doi: 10.1016/j.ygyno.2006.06.025. Epub 2006 Jul 27. PMID 16875720
- [Result] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Result] du Bois A, Reuss A, Pujade-Lauraine E, Harter P, Ray-Coquard I, Pfisterer J. Role of surgical outcome as prognostic factor in advanced epithelial ovarian cancer: a combined exploratory analysis of 3 prospectively randomized phase 3 multicenter trials: by the Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom (AGO-OVAR) and the Groupe d'Investigateurs Nationaux Pour les Etudes des Cancers de l'Ovaire (GINECO). Cancer. 2009 Mar 15;115(6):1234-44. doi: 10.1002/cncr.24149. PMID 19189349
- [Result] Eisenkop SM, Spirtos NM, Friedman RL, Lin WC, Pisani AL, Perticucci S. Relative influences of tumor volume before surgery and the cytoreductive outcome on survival for patients with advanced ovarian cancer: a prospective study. Gynecol Oncol. 2003 Aug;90(2):390-6. doi: 10.1016/s0090-8258(03)00278-6. PMID 12893206
- [Result] Chi DS, Franklin CC, Levine DA, Akselrod F, Sabbatini P, Jarnagin WR, DeMatteo R, Poynor EA, Abu-Rustum NR, Barakat RR. Improved optimal cytoreduction rates for stages IIIC and IV epithelial ovarian, fallopian tube, and primary peritoneal cancer: a change in surgical approach. Gynecol Oncol. 2004 Sep;94(3):650-4. doi: 10.1016/j.ygyno.2004.01.029. PMID 15350354
- [Result] Chi DS, Eisenhauer EL, Zivanovic O, Sonoda Y, Abu-Rustum NR, Levine DA, Guile MW, Bristow RE, Aghajanian C, Barakat RR. Improved progression-free and overall survival in advanced ovarian cancer as a result of a change in surgical paradigm. Gynecol Oncol. 2009 Jul;114(1):26-31. doi: 10.1016/j.ygyno.2009.03.018. Epub 2009 Apr 23. PMID 19395008
- [Result] Chi DS, Zivanovic O, Levinson KL, Kolev V, Huh J, Dottino J, Gardner GJ, Leitao MM Jr, Levine DA, Sonoda Y, Abu-Rustum NR, Brown CL, Barakat RR. The incidence of major complications after the performance of extensive upper abdominal surgical procedures during primary cytoreduction of advanced ovarian, tubal, and peritoneal carcinomas. Gynecol Oncol. 2010 Oct;119(1):38-42. doi: 10.1016/j.ygyno.2010.05.031. Epub 2010 Jul 6. PMID 20609464
- [Result] Schulman-Green D, Ercolano E, Dowd M, Schwartz P, McCorkle R. Quality of life among women after surgery for ovarian cancer. Palliat Support Care. 2008 Sep;6(3):239-47. doi: 10.1017/S1478951508000497. PMID 18662417
- Available data/document: Individual Participant Data Set — https://www.iuct-oncopole.fr/recherches-necessitant-une-reutilisation-de-donnees — All the information is provided on this web page in accordance with the RGPD regulations